CLINICAL TRIAL: NCT06435871
Title: Developing Inclusive Support and Intervention for Spanish-speaking Latiné Prostate Cancer Survivors: Understanding Cultural Nuances in Survivorship Decision Making
Brief Title: Developing Inclusive Support and Intervention for Spanish-speaking Latiné Prostate Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE9824
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Latinos
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cancer treatment outcomes (Experimental): The study population will be divided into three cohorts:
  * Spanish-speaking preferred Latiné,
  * English-speaking preferred Latiné,
  * English-speaking non-Latiné patients.
  Domain assessments between groups will be made using ANOVA with pairwise comparisons.
  Interventions: Behavioral: Expanded Prostate Cancer Index Composite and Decision Regret Scale

INTERVENTIONS:
Behavioral: Expanded Prostate Cancer Index Composite and Decision Regret Scale — This comprehensive instrument measures urinary, sexual, and bowel symptoms in men treated for prostate cancer. It can provide a detailed view of the patient's quality of life post-treatment.

SUMMARY:
Prostate cancer is a significant concern for Latiné men, with over 17,000 new cases annually. Decision-making for treatment is complex, especially due to barriers like low health literacy and cultural factors. Research on survivorship and post-treatment issues like erectile dysfunction is lacking. To improve care, a study will engage 288 participants across various medical facilities, including 100 at Cleveland Clinic. Thirty subjects will participate in focus groups representing Spanish-speaking Latiné, bilingual Latiné, and English-speaking non-Latiné individuals to understand their perspectives and enhance communication. This aims to develop tailored resources, like Spanish-language educational videos, addressing language and cultural needs for informed decision-making.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-skin cancer among Latiné men, with over 17,000 new cases yearly. While most men live with the disease rather than die from it, ensuring quality of life is crucial in treatment decisions. Latiné men face unique decision-making challenges due to low health literacy, barriers to healthcare access, and cultural differences in treatment understanding and communication. Decision aids that consider patient values and cultural nuances like familismo are essential for effective shared decision-making.

Despite the significance of racial and ethnic disparities in prostate cancer outcomes, research has been limited, especially among Latiné populations. The CEASAR study highlighted the need for more inclusive research, showing no significant outcome differences across racial groups but underrepresenting Latiné men. The Urology Care Foundation has provided Spanish-language resources, yet there's a gap in materials discussing treatment choices in the context of sexual, bowel and urinary health post-treatment.

This gap underlines the necessity for research focused on the Latiné community's perspectives on prostate cancer survivorship, particularly concerning erectile dysfunction, bowel function and urinary function. This study aims to fill this void through focus groups to better understand Latiné men's views and enhance patient education and shared decision-making. A Spanish-language educational video informed by these insights will address the critical need for culturally and linguistically appropriate resources, bridging the information gap for Spanish-speaking survivors

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Diagnosis of Localized Prostate Cancer
* Underwent radical prostatectomy by their urological surgeon
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patient whose primary language is not English or Spanish
* Patients who had brachytherapy and/or radiation treatment as their initial treatment
* Patients with disease progression at time study recruitment who are requiring other treatments (ADT, chemotherapy, immunotherapy)
* Patients who underwent current non-standard prior treatment options for localized prostate cancer including cryotherapy and high intensity focused ultrasound (HIFU)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Urinary health-related QoL as measured using the validated EPIC-26 questionnaire | During group interview (minimum of three 90-minute sessions) post radical prostatectomy
  The EPIC questionnaire evaluates urinary health-related quality of life domains specific to prostate cancer patients: It is a 13-question survey, where 1-5 are focused on the urinary health. Responses are given on a Likert scale, ranging from "very poor" to "very good" or "no problem" to "big problem," depending on the question.One-way ANOVA test is used for comparison of EPIC domains between the three cohorts.
Bowel health-related QoL as measured using the validated EPIC-26 questionnaire | During group interview (minimum of three 90-minute sessions) post radical prostatectomy
  The EPIC questionnaire evaluates bowel health-related quality of life domains specific to prostate cancer patients: It is a 13-question survey, where questions 6-7 are focused on the bowel health. Responses are given on a Likert scale, ranging from "very poor" to "very good" or "no problem" to "big problem," depending on the question.One-way ANOVA test is used for comparison of EPIC domains between the three cohorts.
Sexual health-related QoL as measured using the validated EPIC-26 questionnaire | During group interview (minimum of three 90-minute sessions) post radical prostatectomy
  The EPIC questionnaire evaluates sexual health-related quality of life domains specific to prostate cancer patients: It is a 13-question survey, where questions 8-12 are focused on the sexual health. Responses are given on a Likert scale, ranging from "very poor" to "very good" or "no problem" to "big problem," depending on the question.One-way ANOVA test is used for comparison of EPIC domains between the three cohorts.
Hormonal health-related QoL as measured using the validated EPIC-26 questionnaire | During group interview (minimum of three 90-minute sessions) post radical prostatectomy
  The EPIC questionnaire evaluates hormonal health-related quality of life domains specific to prostate cancer patients: It is a 13-question survey, where question 13 is focused on the hormonal health. Responses are given on a Likert scale, ranging from "very poor" to "very good" or "no problem" to "big problem," depending on the question.One-way ANOVA test is used for comparison of EPIC domains between the three cohorts.
QoL as measured using the combined score of EPIC-26 questionnaire | During group interview (minimum of three 90-minute sessions) post radical prostatectomy
  The EPIC questionnaire evaluates health-related quality of life domains specific to prostate cancer patients: It is a 13-question survey. Responses are given on a Likert scale, ranging from "very poor" to "very good" or "no problem" to "big problem," depending on the question.One-way ANOVA test is used for comparison of EPIC domains between the three cohorts.

SECONDARY OUTCOMES:
Decisional conflict as assesed by decisional conflict scores | During group interview (minimum of three 90-minute sessions) post radical prostatectomy
  The DRS is a 5-item Likert scale with responses ranging from 1 (strongly agree) to 5 (strongly disagree), designed to evaluate distress or remorse following a healthcare decision. Comparison of decisional conflict scores between the study groups using one-way ANOVA testing.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Weight, MD, Principal Investigator — Cleveland Clinic Glickman Urological and Kidney Institute, Cleveland Clinic Foundation, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Glickman Urological and Kidney Institute, Cleveland Clinic Foundation, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for the duration of the study ~ 2 years.
Access Criteria: Each institution will collect their own patient data into their own RedCap. No PHI data will be shared amongst the institutions - only de-identified data will be shared from CCF to UCSD via REDCAP and included in analyses which will be performed by specialist data analysts at UCSD and by investigators listed on this IRB. Access to the data will be limited to authorized personnel only, who will be required to maintain strict confidentiality and adhere to data protection regulations.